CLINICAL TRIAL: NCT00947154
Title: Open Label Trial of Aripiprazole in Trichotillomania.
Brief Title: Trial of Aripiprazole in Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lorrin M Koran, Professor or Psychiatry, Emeritus, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-07172009-3320; eProtocol #15291 (Other Grant/Funding Number: NIMH T32 training grant)
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Results first posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-05

CONDITIONS: Trichotillomania
Keywords: trichotillomania; aripiprazole; treatment
MeSH Terms: conditions — Trichotillomania | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label aripiprazol (Experimental): Aripiprazole dose of 5 mg/d, which could be reduced to 2 mg/d if the initial dose was not tolerated. Dose was increased by up to 5 mg at intervals of 2 weeks until a maximum target dosage of 15 mg/d was reached at the beginning of week 5. Dose was not increased if the subject showed clinical improvement at a lower dose, defined as a 50% reduction in Massachusetts General Hospital Hair Pulling Scale (MGHHPS), or was intolerant of a further dosing increase. Dose was not increased after week 5; at any point, it could be decreased secondary to side effects.
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: aripiprazole — aripiprazole dose of 5 mg/d, which could be reduced to 2 mg/d if the initial dose was not tolerated. Dose was increased by up to 5 mg at intervals of 2 weeks until a maximum target dosage of 15 mg/d was reached at the beginning of week 5. Dose was not increased if the subject showed clinical improvement at a lower dose, defined as a 50% reduction in Massachusetts General Hospital Hair Pulling Scale (MGHHPS), or was intolerant of a further dosing increase. Dose was not increased after week 5; at any point, it could be decreased secondary to side effects.
  Other Names: Abilify

SUMMARY:
No medication has been reliably shown to benefit those suffering from trichotillomania (compulsive hair pulling). The current study proposes to evaluate the effectiveness of the medication aripiprazole for treatment of trichotillomania (TTM). Patients will take a gradually increased dose of the medication in an open-label study to see whether it relieves hair-pulling urges, decreases hair pulling behavior and is well tolerated.

DETAILED DESCRIPTION:
The proposed study is an 8-week, open-label trial of aripiprazole. The study would enroll 10 patients diagnosed with TTM meeting DSM-IV criteria. Subjects would start at a dose of 5 mg, which can be reduced to 2 mg if initial dose is not tolerated. Dose will be increased by 5 mg every two weeks (or as tolerated, with a minimum increase of 2 mg) until a maximum target dose of 15 mg is reached at the beginning of week 5. Dosing would not be increased if a patient showed clinical improvement at a lower dose (defined as a 30% reduction in Massachusetts General Hairpulling Scale) or was intolerant of a further dose increase. Dose may not be increased after week 5; at any point it may be decreased because of intolerability. Modified dosing of aripiprazole will not automatically happen if a patient is taking fluoxetine or paroxetine, but awareness that increased aripiprazole levels are associated with P450 2D inhibition (and consequent tolerability of a given dose) may factor into clinical decisions to increase, maintain or decrease aripiprazole dosage.

Effectiveness: The primary measure of drug effect would be a change from baseline to endpoint in the Massachusetts General Hospital Hairpulling Scale (MGHHS) as well as the actual-pulling subscale (items 4,5,6; MGHHS-AP). Secondary measures would include the Clinical Global Impressions_Improvement scale (CGI-I), 17-item Hamilton Depression Scale (HAM-D) and the Hamilton Anxiety Scale (HAM-A).

Assessments: Primary efficacy measures will be assessed at baseline and at the end of weeks 2, 4, 6 and 8, or early termination. Week 2 and 6 follow-ups may occur over the telephone. Safety and tolerability will be assessed at each two-week interval. Secondary end-points will be assessed at baseline and weeks 4 and 8, or early termination.

Type and Number of Experimental Subjects and Controls: This study would enroll 10 patients at Stanford in a single-site study. Inclusion and exclusion criteria are described separately. Children will not be included in this proposed study, because the Investigator does not have clinical competency in child psychiatry and childhood Trichotillomania may be a different disorder than the condition seen in adults.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients:

* Must be outpatients between the ages of 18 and 65 at the start of study
* May be male or female
* Have DSM-IV trichotillomania of at least 6 months duration
* Allowed psychotropic medications are limited to:

  * SSRIs (citalopram, escitalopram, fluoxetine, fluvoxamine, paroxetine, sertraline), SNRIs (duloxetine, venlafaxine) and mirtazapine, as long as the dosage has not changed for 4 weeks prior to study enrollment.
  * Other allowed medications include non-hypnotic sleeping agents, specifically trazodone, diphenhydramine, hydoxyzine and ramelteon.
  * If a patient is taking non-allowed psychotropic medications, he/she must be titrated off by the prescribing physician and be off of the medication for at least 2 weeks prior to trial enrollment.
* We will not exclude patients meeting DSM-IV criteria for:

  * body dysmorphic disorder;
  * major depression;
  * dysthymia;
  * GAD, social phobia, panic disorder.

Exclusion Criteria:

* We will exclude patients suffering from:

  * organic mental disorders;
  * psychotic mental disorders including delusional disorder, somatic type;
  * mental retardation or developmental disabilities;
  * substance or alcohol abuse;
  * depressive disorders with current suicidal risk;
  * factitious disorders;
  * dissociative disorders;
  * obsessive compulsive disorder;
  * personality disorders sufficiently severe to interfere with cooperation with the study;
  * bipolar I or II disorder.
* Patients taking psychotropic agents other than those specifically listed in item d above. If a patient is taking non-allowed psychotropic medications, he/she must be titrated off such medications by the prescribing physician and be off of the medication for 2 weeks prior to trial enrollment.
* Pregnant or nursing women.
* Patients with a known hypersensitivity or allergy to aripiprazole.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorrin M Koran, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] White MP, Koran LM. Open-label trial of aripiprazole in the treatment of trichotillomania. J Clin Psychopharmacol. 2011 Aug;31(4):503-6. doi: 10.1097/JCP.0b013e318221b1ba. PMID 21694623

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Aripiprazol: Aripiprazole dose of 5 mg/d could be reduced to 2 mg/d if initial dose not tolerated. Dose increased by up to 5 mg q 2 weeks to max dose of 15 mg/d at start of week 5. Dose not increased if subject showed clinical improvement at a lower dose, defined as 50% decrease in Mass General Hospital Hair Pulling Scale (MGHHPS), or was intolerant of dosing increase. Dose not increased after week 5; at any point, it could be decreased for side effects.
Period: Overall Study
Arm/Group | Open-label Aripiprazol
Started | 12
Completed | 11
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Aripiprazol
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mass General Hair Pulling Scale
Description: A brief, self-report instrument for assessing repetitive hairpulling. Seven individual items, rated for severity from 0 to 4, assess frequency and intensity of urges to pull, ability to control the urges, frequency of pulling, attempts to resist pulling, success in resisting, and associated distress. Statistical analyses indicate that the seven items form a homogenous scale for the measurement of severity in trichotillomania. Higher scores indicate greater severity of hair pulling. Total score can range from 0 to 28.
Time Frame: Change from baseline to week 8
Population: 11 of the 12 subjects initially enrolled. One was lost to follow-up after baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Aripiprazol
Number analyzed (Participants) | 11
units on a scale | -7.8 (7.8)

2. Secondary Outcome: CGI-I Score of 1 or 2 (Very Much or Much Improved)
Description: CGI = Clinical Global Improvement 7-item scale, from very much worse to very much better.
Time Frame: At week 8
Population: 11 of the 12 subjects initially enrolled. One subject was lost to follow-up after the baseline visit.
Measure: Number; unit: participants
Arm/Group | Open-label Aripiprazol
Number analyzed (Participants) | 11
participants | 7

3. Primary Outcome: Mass General Hair Pulling Scale, Actual Pulling Subscale
Description: Sum of scores for items 4, 5 and 6 from the Mass General Hair Pulling Scale (Frequency of Pulling, Attempts to Resist Pulling, Control Over Hair Pulling). Score can range from 0 to 12; higher scores indicate more severe hair pulling.
Time Frame: change from baseline to end of week 8
Population: 11 participants. 1 participant was lost to follow-up after week 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Aripiprazol
Number analyzed (Participants) | 11
units on a scale | -3.9 (4.1)

4. Secondary Outcome: Clinical Global Impressions Improvement (CGI-I)
Description: The CGI-I is a clinician rated scale ranging from 0 (not assessed) to 7 (very much worse), with intermediate scores of 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse). The clinician is rating the overall change in the patient's clinical condition.
Time Frame: At week 8
Population: 11 participants. 1 participant lost to follow up after week 1
Measure: Number; unit: percentage completers with score 1 or 2
Arm/Group | Open-label Aripiprazol
Number analyzed (Participants) | 11
percentage completers with score 1 or 2 | 64

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: In-person visits at baseline, and weeks 4 and 8. A telephone check-in was performed at weeks 2 and 6.
Arm/Group | Open-label Aripiprazol
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Aripiprazol (N=11)
akathisia (Nervous system disorders) | 6
insomnia (Psychiatric disorders) | 4
anxiety (Psychiatric disorders) | 4
dry mouth (Gastrointestinal disorders) | 3
blurry vision (Eye disorders) | 3
dizziness (Nervous system disorders) | 2
anorgasmia (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No